CLINICAL TRIAL: NCT07381114
Title: Phase II Clinical Study on the Efficacy and Safety of Ivarmacitinib in Preventing Acute Graft-versus-host Disease After HLA-matched Transplantation
Brief Title: A Clinical Study on the Efficacy and Safety of Ivarmacitinib in Preventing aGVHD After HLA-matched Transplantation
Acronym: Ivarmacitinib
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT2025130
Record Dates: First submitted 2025-11-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: aGVHD
Keywords: Ivarmacitinib; aGVHD
MeSH Terms: interventions — ivarmacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivarmacitinib (Experimental): During the dose exploration phase, the "3+3" method was used for Ivarmacitinib, with the dose incrementing from 2mg to 6mg. The medication was administered starting from -3 days and observation continued until 28 days after transplantation to determine the RP2D dose. Patients at the RP2D dose during the dose exploration phase were enrolled in the expansion study. Patients in the expansion study received RP2D Ivarmacitinib treatment daily for 3 days to 100 days.
  Interventions: Drug: Ivarmacitinib

INTERVENTIONS:
Drug: Ivarmacitinib — Patients at the RP2D dose during the dose exploration phase were enrolled in the expansion study. Patients in the expansion study received RP2D Ivarmacitinib treatment daily for 3 days to 100 days.

SUMMARY:
To apply Ivarmacitinib for the prevention of acute graft-versus-host disease (aGVHD) in HLA haploidentical transplantation, the incidence of grade II-IV aGVHD after prevention, the incidence of primary graft failure, the rate of GVHD-free relapse-free survival (GRFS) (12 months), the incidence of infection, the incidence of chronic graft-versus-host disease (cGvHD) (100 days - 1 year), treatment-related mortality, the incidence and severity of cytokine release syndrome (CRS), and the safety of the prevention regimen will be evaluated.

DETAILED DESCRIPTION:
This project is a prospective, single-arm clinical study. It aims to apply Ivarmacitinib for the prevention of acute graft-versus-host disease (aGVHD) in patients with hematological malignancies undergoing HLA-mismatched transplantation. The primary objective is to observe the incidence of grade II-IV aGVHD after transplantation prevention. The secondary objectives include the incidence of primary graft failure, graft-versus-host disease-free and relapse-free survival (GRFS) at 12 months, the incidence of infection, the incidence of chronic graft-versus-host disease (cGvHD) within 100 days to 1 year, treatment-related mortality, the incidence and severity of cytokine release syndrome (CRS), and the safety assessment of the prevention regimen. This study is intended to provide a reference for the clinical application of Ivarmacitinib in transplantation. Therefore, this research is proposed to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* The patients have been clearly diagnosed with hematological malignancies, including acute myeloid leukemia, acute lymphocytic leukemia, chronic myeloid leukemia, myelodysplastic syndrome, non-Hodgkin's lymphoma, and Hodgkin's lymphoma. The planned treatment for these patients is myeloablative or reduced-intensity conditioning, followed by HLA half-matched stem cell transplantation.
* Has not received any systemic treatment, including extracorporeal photodynamic therapy (ECP)
* KPS>60% or ECOG PS 0-2
* Patients who have not received any other prophylactic immunosuppressive agents or aGVHD/cGVHD treatment are eligible
* The female subjects of childbearing age are willing to use a medically approved highly effective contraceptive method (such as intrauterine device, contraceptive pill or condom) during the study period and within 180 days after the last administration of the study drug; for male subjects whose partners are of childbearing age, they agree to use an effective contraceptive method during the study period and within 180 days after the last administration of the study drug

Exclusion Criteria:

* Pregnant women or women who are breastfeeding
* Absolute Neutrophil Count (ANC) < 1.0 x 109/L or Platelet Count < 50 x 109/L
* Uncontrolled active infections or active hepatitis B or hepatitis that requires antiviral treatment
* Human Immunodeficiency Virus (HIV) positive
* Uncontrolled concurrent diseases, including but not limited to persistent or active infections, autoimmune diseases, thrombosis, symptomatic congestive heart failure, unstable angina pectoris, unstable arrhythmias, or mental disorders/situations that would limit compliance with the study requirements
* There are severe respiratory system diseases, severe renal function impairment, clinically significant or uncontrolled heart diseases, unresolved cholestasis and liver diseases (not attributable to aGvHD). Diseases that interfere with coagulation or platelet function and/or current drug treatments
* Immunosuppressive doses of steroids. This does not exclude the use of steroids in subjects with adrenal cortical insufficiency
* The diagnosis was clear: chronic lymphocytic leukemia, marginal zone lymphoma (MALT type), smoldering multiple myeloma, etc., all being low-grade malignant/cancer-preventing blood tumors
* Patients who have been diagnosed with pre-transplantation digestive tract perforation and have a history of gastric or intestinal resection surgeries, etc., may have their drug absorption affected
* It is known that there may be allergic reactions, hypersensitivity reactions or intolerance to the studied drug or its excipients
* The researchers believe that there are any conditions that might harm the subjects or prevent them from fulfilling or meeting the requirements of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of grade II-IV aGVHD | up to 2 years

SECONDARY OUTCOMES:
the incidence of primary graft failure | up to 2 years
the event-free survival (GRFS) without GVHD (12 months) | 12 months